CLINICAL TRIAL: NCT03499106
Title: An Open-label, 2-Period, Fixed-sequence, Phase 1 Study in Healthy Volunteers to Evaluate the Effect of Itraconazole, a Potent CYP3A Inhibitor, on the Pharmacokinetics of IW-1973
Brief Title: A Trial to Evaluate the Effect of Itraconazole (ITZ), a CYP3A4 Inhibitor, on the Pharmacokinetics of Praliciguat (IW-1973) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cyclerion Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: C1973-104
Record Dates: First submitted 2018-04-09; First posted 2018-04-17 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Healthy
MeSH Terms: interventions — praliciguat; Itraconazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Healthy Volunteers (Experimental): Period 1: Single dose of IW-1973. Period 2: ITZ is dosed once daily (QD) for 17 days; a single dose of IW-1973 is administered 1 hour after the fourth ITZ QD dose.
  Interventions: Drug: IW-1973; Drug: Itraconazole

INTERVENTIONS:
Drug: IW-1973 — Oral Tablet
Drug: Itraconazole — Oral Capsule

SUMMARY:
The primary objective of the study is to evaluate the effect of itraconazole (a potent cytochrome P450 isoenzyme [CYP]3A inhibitor) on the pharmacokinetics of IW-1973.

ELIGIBILITY:
Inclusion Criteria:

* Subject is an ambulatory adult between 18 and 75 years old at the screening visit
* Subject is in good health and has no clinically significant findings on physical examination
* Body mass index is > 18 and < 30.0 kg/m2 at the screening visit
* Women of reproductive potential must have a negative pregnancy test at the time of check-in and must agree to use protocol-specified contraception throughout the duration of the study and for 2 months after the final dose of study drug
* Men must agree to use protocol-specified contraception and also to not donate sperm throughout the study and for 2 months after the final dose of study drug
* Other inclusion criteria per protocol

Exclusion Criteria:

* Any active or unstable clinically significant medical condition
* Use of any prescribed or non-prescribed medication
* Other exclusion criteria per protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-04-12 (Actual); Primary Completion 2018-07-06 (Actual); Study Completion 2018-07-06 (Actual)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration Time Curve of IW-1973 From Time Zero Extrapolated to Infinity (AUC[0-inf]) | Predose and up to 14 days post dose of IW-1973
Maximum Observed Plasma Concentration (Cmax) of IW-1973 | Predose and up to 14 days post dose of IW-1973

SECONDARY OUTCOMES:
Time to Cmax (Tmax) of IW-1973 | Predose and up to 14 days post dose of IW-1973
Area Under the Concentration-Time Curve From Time Zero to 24 hours AUC(0-24) Postdose of IW-1973 | Predose and up to 14 days post dose of IW-1973
Area Under the Concentration-Time Curve From Time Zero to Time of Last Quantifiable Concentration (AUC[0-last]) of IW-1973 | Predose and up to 14 days post dose of IW-1973
Apparent Terminal Half-Life (t1/2) of IW-1973 | Predose and up to 14 days post dose of IW-1973
Apparent Terminal Rate Constant (lambda[z]) of IW-1973 | Predose and up to 14 days post dose of IW-1973
Apparent Total Plasma Clearance (CL/F) of IW-1973 | Predose and up to 14 days post dose of IW-1973
Apparent Volume of Distribution (Vz/F) of IW-1973 | Predose and up to 14 days post dose of IW-1973

CONTACTS AND LOCATIONS:
Locations (1):
- IQVIA, Overland Park, Kansas, United States